CLINICAL TRIAL: NCT01455636
Title: Preventing Linear Growth Faltering and Reversal of Stunting Among Low Birth Weight Infants in Bangladesh: a Community-based Cluster Randomized Control Trial
Brief Title: Preventing Linear Growth Faltering Among Low Birth Weight Infants in Bangladesh
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Stanley Zlotkin, Chief, Global Child Health, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1000014576
Record Dates: First submitted 2011-10-16; First posted 2011-10-20 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Infant, Low Birth Weight
Keywords: pediatric; micronutrient powder; hand hygiene; low birth weight; infant feeding; hand sanitizers
MeSH Terms: interventions — Hand Sanitizers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hand hygiene with Hand Sanitizer (HS) (Experimental): To obtain 480 low birth weight infants the entire area of Kaliganj and Norsinghdi will be divided into 48 clusters based on the list of pregnant women identified through a household survey.
  24 clusters will be randomized to receive Hand Sanitizer plus nutrition and hygiene education and the remaining 24 will receive only nutrition and hygiene education.
  Interventions: Other: Hand Sanitizer
- Hand hygiene with no Hand Sanitizer (Experimental): To obtain 480 low birth weight infants the entire area of Kaliganj and Norsinghdi will be divided into 48 clusters based on the list of pregnant women identified through a household survey.
  24 clusters will be randomized to receive Hand Sanitizer plus nutrition and hygiene education and the remaining 24 will receive only nutrition and hygiene education.
  Interventions: Other: Hand Sanitizer; Dietary Supplement: Improved Micronutrient Powder
- Micronutrient Powder (Experimental): From 6 months of age, children in randomized clusters will be assigned to receive one sachet of Improved Micronutrient Powder, I-MNP per day for six months with or without hand sanitizer.
  Throughout the entire intervention period, mothers/caregivers of the children in all groups will receive simple, standardized, and age and culturally appropriate nutrition and health education that aims to improve feeding and health-seeking behavior and caring practices.
  Interventions: Dietary Supplement: Improved Micronutrient Powder; Dietary Supplement: No Micronutrient Powder
- Control (Placebo Comparator): From 6 months of age, children in randomized clusters will be assigned to receive no hand sanitizer or no micronutrient powder
  Throughout the entire intervention period, mothers/caregivers of the children in all groups will receive simple, standardized, and age and culturally appropriate nutrition and health education that aims to improve feeding and health-seeking behavior and caring practices.
  Interventions: Other: No hand sanitizer; Dietary Supplement: No Micronutrient Powder

INTERVENTIONS:
Other: Hand Sanitizer — The water-based hand sanitizer to be used in the current project will be produced in India by Hexagon Inc. It will be dispensed via a foam dispenser, since it has been established that foam is preferable to gel because of the natural tendency to rub foam more thoroughly into one's hands.
  Arms: Hand hygiene with Hand Sanitizer (HS); Hand hygiene with no Hand Sanitizer
Dietary Supplement: Improved Micronutrient Powder — A modified and improved formulation of MNPs will be used. The composition is specially designed to enhance appetite and growth with 17 essential micronutrients; including calcium and magnesium, as well as an increased amount of zinc (10 mg). Previously MNP formulations (including the UNICEF formulation) contained only 5 mg of zinc and did not contain magnesium and calcium, which are essential nutrients for bone formation.
  Other Names: MNP
  Arms: Hand hygiene with no Hand Sanitizer; Micronutrient Powder
Other: No hand sanitizer — All family members will receive hand-hygiene education with Information, Education and Communication (IEC) materials including pictorial messages describing critical points for hand-hygiene.
  No placebo for the hand sanitizers will be provided to families in Groups 3 and 4 because it would be unethical if families were to use an inactive hand-hygiene product as a substitute for routine hand-washing. Nevertheless, all groups will be instructed
  Arms: Control
Dietary Supplement: No Micronutrient Powder — I-MNP and placebo will be procured from a local pharmaceutical company in Dhaka, Bangladesh (Renata Pharma Ltd.). The outer-packaging of the sachets of 'I-MNP' and 'placebo-MNP' will be identical except for a different numeric code for each.
  Arms: Control; Micronutrient Powder

SUMMARY:
Low birth weight (LBW) infants are particularly vulnerable to frequent infections and consequent morbidity resulting in sub-optimal breastfeeding, limited ingestion of complementary foods and ultimately micronutrient deficiencies that result in post-natal linear growth faltering. The objective of this study is to facilitate improved feeding practices through the early reduction of infections using the innovative tools of water-based hand sanitizer (beginning at birth) and an improved micronutrient powder (I-MNP) (beginning at 6 months of age). A community-based cluster randomized controlled trial will be carried out in Bangladesh using a 2x2 factorial design. LBW infants (n=480) will be recruited at birth and allocated to either HS or No HS from 0 to 6 months. From 6 to 12 months, half of the children in each group will be randomized to receive I-MNP. All groups will receive nutrition and hygiene education from birth to 12 months. Recumbent length is the primary outcome; morbidity, dietary intake and hemoglobin will be assessed as secondary outcomes. By working with BRAC, the largest implementation agency in Bangladesh, there is the opportunity to translate the results directly and quickly into child health programs in Bangladesh.

DETAILED DESCRIPTION:
General Objective To explore the relative effect of hand sanitizer and home fortification with an improved MNP (plus nutrition education) to prevent infections, improve feeding and ultimately to improve growth among LBW infants in Bangladesh.

Specific Objectives Although the applicants clearly understand that the primary purpose of the Alive and Thrive RFP is to improve infant feeding, we believe that by preventing infections, feeding will improve and growth will accelerate. Thus our primary objective is to determine the relative effect of intervention packages to improve feeding and thus prevent or reverse linear growth faltering and reduce rates of stunting among LBW infants (Ha: Combination of all three interventions will improve feeding and prevent or reverse linear growth faltering and reduce rates of stunting)

Secondary objectives (i) Investigate the effect of intervention packages on rates of diarrhea and acute respiratory tract infection (ARI).

(Ha: Combination of all three interventions will reduce on rates of diarrhea and acute respiratory tract infection) (ii) Explore the effect of the intervention packages on energy and nutrient intakes of infants and their feeding behaviors.

(Ha: Combination of all three interventions will increase energy and nutrient intakes of infants and improve the feeding behaviors) (iii) Determine the impact of the improved MNP on iron status (hemoglobin level in blood) in a subgroup.

(Ha: The group receiving the improved MNP will have increased hemoglobin level in blood and reduced rates of anemia)

ELIGIBILITY:
Inclusion Criteria:

* infants born as singletons and full term (mothers will be identified at ~8 months or >37 weeks gestation to avoid including premature babies who are at high risk of neonatal mortality).
* must have a birth weight ≥1800g and <2500g.
* Families involved in the study must be planning to remain in the study community for the next 12 months
* written consent must be received from an authorized guardian.
* all pregnant women will be identified and visited during their 8th month of pregnancy. A local informant will be identified for birth notification, who will inform the CHW (with a cell phone) when a child is born. All newborns will be screened and those who meet the inclusion criteria will be enrolled.

Exclusion Criteria:

* newborns with severe illnesses or congenital abnormalities /severe malformations that affect feeding will be excluded from the study.
* infants whose mothers did not survive during childbirth will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Anthropometry - Recumbent Length | Change from baseline in length over 12 months
  Recumbent length will be measured to 0.01cm on a locally constructed wooden stadiometer. Anthropometric data will be converted to Z-scores using the WHO growth standards.
Anthropometry - Weight | Change from baseline in weight over 12 months
  weight using an infant balance with 15 g precision (SECA Model 345) calibrated on a regular, scheduled basis. Anthropometric data will be converted to Z-scores using the WHO growth standards.

SECONDARY OUTCOMES:
Infectious Morbidity | Weekly for 52 weeks
  Diarrhea will be defined as >3 loose stools in a 24-h period or >1 loose stool containing blood. Mothers are expected to use ORS and zinc tablets for all diarrhea episodes (provided free to study subjects irrespective of study group). Acute Respiratory Infections (ARI) will be diagnosed according to World Health Organization Criteria Information on the occurrence, type and severity of diarrhea and ARI and health seeking be collected weekly.
Infant and young child feeding | Monthly for 12 months
  Information on age-specific feeding practices will be obtained monthly by trained nutritionists using standardized infant and young child feeding indicators.
Blood collection and Hemoglobin (Hb) measurement | 6 and 12 months post randomization
  A standardized finger-prick technique will be used to collect blood from the infants from a subsample of Groups 2 and 4 (at 6 and 12 months). Hb will be measured using a portable Hemocue (Hemocue Inc.).
Socioeconomic status (SES) and demographic information | Baseline
  Household SES will be assessed by a pre-coded structured interview designed to obtain information on the household demographic structure, parental education, employment, material possessions and by inspection of housing quality.
Household Food Security | Baseline
  Information on household food security will be collected using standardized questionnaires used in the same population.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Zlotkin, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Research and Evaluation Division, BRAC, Dhaka, Bangladesh
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Shafique S, Sellen DW, Lou W, Jalal CS, Jolly SP, Zlotkin SH. Mineral- and vitamin-enhanced micronutrient powder reduces stunting in full-term low-birth-weight infants receiving nutrition, health, and hygiene education: a 2 x 2 factorial, cluster-randomized trial in Bangladesh. Am J Clin Nutr. 2016 May;103(5):1357-69. doi: 10.3945/ajcn.115.117770. Epub 2016 Apr 6. PMID 27053383
- [Derived] Singla DR, Shafique S, Zlotkin SH, Aboud FE. A 22-element micronutrient powder benefits language but not cognition in Bangladeshi full-term low-birth-weight children. J Nutr. 2014 Nov;144(11):1803-10. doi: 10.3945/jn.114.193094. Epub 2014 Aug 20. PMID 25143374